CLINICAL TRIAL: NCT05423782
Title: Prevalence of Mental Disorder and Somatic Co-morbidities Among Asylum Seekers in Marseille
Acronym: PREMENTADA
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM20_0196
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Global Health of Asylum Seekers in France

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction : World Health Organization (WHO) considers that the heterogeneity of concepts and definitions of migrants is an obstacle to obtaining evidence to inform public health policies. Thus, it recommends distinguishing refugees from asylum seekers. Asylum seekers are migrants who recently arrived in their host country and whose administrative situation is being examined. They do not have the same access to health care or the same rights as refugees.

In France in 2021, 78,372 major people filled a first asylum application, a 26.4% increase compared to 2020 Regarding the mental health of exiles, a literature review informs us that 31.5% of them suffer from post-traumatic stress disorder (PTSD), 31.5% from depression and 11.1% from anxiety disorders. However, these data are taken from studies that do not make a distinction between refugees and asylum seekers These missing data are a hindrance to the development of efficient strategies for the management of these populations within the health systems of Western countries.

The primary objective of this study was to describe the health status of asylum seekers who have recently arrived in their Western host country. The secondary objective was to investigate potential explanatory factors for the health status of asylum seekers.

Method: Single-center, cross-sectional, observational epidemiological study. The Refugee health screener (RHS15) questionnaire and the Cumulative Illness Rating Scale (CIRS) will be administered by a trained interviewer to each patient included on the day of their inclusion, in the asylum seekers reception platform (PADA).Potential use of tobacco, existence of an adapted treatment in case of a detected pathology and certain socio-demographic data will also be collected.

A telephone interpreting service will be used in the case of an allophone patient whose spoken language is not spoken by the interviewer. Each patient included will have an appointment to perform a standardised blood and urine sample.

Benefits : PREMENTADA study will provide a better understanding of the health status of the population of asylum seekers in France. As the existence of data is a prerequisite for evidence-based medicine, we notice the lack of previous studies specifically addressing this population in France.

DETAILED DESCRIPTION:
Introduction : World Health Organization (WHO) considers that the heterogeneity of concepts and definitions of migrants is an obstacle to obtaining evidence to inform public health policies. Thus, it recommends distinguishing refugees from asylum seekers. Asylum seekers are migrants who recently arrived in their host country and whose administrative situation is being examined. They do not have the same access to health care or the same rights as refugees.

In France in 2021, 78,372 major people filled a first asylum application, a 26.4% increase compared to 2020 Regarding the mental health of exiles, a literature review informs us that 31.5% of them suffer from post-traumatic stress disorder (PTSD), 31.5% from depression and 11.1% from anxiety disorders. However, these data are taken from studies that do not make a distinction between refugees and asylum seekers These missing data are a hindrance to the development of efficient strategies for the management of these populations within the health systems of Western countries.

The primary objective of this study was to describe the health status of asylum seekers who have recently arrived in their Western host country. The secondary objective was to investigate potential explanatory factors for the health status of asylum seekers.

Method: Single-center, cross-sectional, observational epidemiological study. The Refugee health screener (RHS15) questionnaire and the Cumulative Illness Rating Scale (CIRS) will be administered by a trained interviewer to each patient included on the day of their inclusion, in the asylum seekers reception platform (PADA).Potential use of tobacco, existence of an adapted treatment in case of a detected pathology and certain socio-demographic data will also be collected.

A telephone interpreting service will be used in the case of an allophone patient whose spoken language is not spoken by the interviewer. Each patient included will have an appointment to perform a standardised blood and urine sample.

Benefits : PREMENTADA study will provide a better understanding of the health status of the population of asylum seekers in France. As the existence of data is a prerequisite for evidence-based medicine, we notice the lack of previous studies specifically addressing this population in France.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Coming to asylum seekers reception platform in Marseille
* Have the cognitive capacity to consent to participation in the study
* Holders of a first asylum application receipt (not older than 21 days )

Exclusion Criteria:

- Existence of cognitive disorders (dementia, mental retardation) or language difficulties (dysphasia, aphasia) limiting understanding and expression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asylum Seekers in France
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Refugee Health Screener (RHS-15) | 30 minutes
  The RHS-15 is a valid 15-item instrument screening to detect on asylum seekers and refugees Post traumatic stress disorder (PTSD), anxiety or depression symptoms. 14 items are rated on a 5-point Likert scale (0 = not at all to 4 = extremely). The last item is assessing the general ability to handle stress on a 5-point Likert scale and a distress thermometer (DT) ranging from 0 to 10. A screening result is positive if the sum of the first 14 items ≥ 12 or if the DT is ≥ 5

SECONDARY OUTCOMES:
Cumulative Illness Rating Scale (CIRS) | 20 minutes
  The CIRS is a comprehensive measure of multimorbidity previously validated on homeless people. Each item is assigned a severity score by means of an assessment of the impact on the patient: 1 (no problem), 2 (current mild problem or past significant problem), 3 (moderate disability or morbidity), 4 (severe problem), 5 (extremely severe or life-threatening problem). The CIRS classifies all items into 14 body systems (including one on mental disorder) to obtain a final cumulative score.

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Khouani J, Jeannu E, Borlot J, Tinland A, Thery D, Jego M, Gentile G, Auquier P, Tabele C. Care pathway of asylum seekers in the health care access points following inclusion in the PREMENTADA project: an observational study. Public Health. 2024 Jul;232:138-145. doi: 10.1016/j.puhe.2024.04.023. Epub 2024 May 22. PMID 38776589